CLINICAL TRIAL: NCT06719622
Title: Evaluation of the Efficacy of Local Budesonide Treatment in Children with Crohn's Disease Located in the Esophagus And/or Stomach And/or Duodenum
Acronym: BETHESDa-CD
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Jagiellonian University (Other); Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABM01
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Crohn Disease (CD)
Keywords: children; esophagus; upper digestive tract; duodenum; stomach; pediatrics; gastroscopy; gastrointestinal endoscopy; local treatment; glucocorticosteroids; omeprazole; proton pump inhibitor
MeSH Terms: conditions — Crohn Disease | interventions — Budesonide; Omeprazole; Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Budesonide (Experimental)
  Interventions: Drug: budesonide
- Omeprazole (Active Comparator)
  Interventions: Drug: omeprazole (proton pump inhibitor)

INTERVENTIONS:
Drug: budesonide — 1 mg budesonide ampoule twice daily for patients weighing ≤35 kg or 2 mg twice daily for patients weighing >35 kg
  Arms: Budesonide
Drug: omeprazole (proton pump inhibitor) — omeprazole 10 mg twice daily for patients weighing ≤35 kg or 20 mg twice daily for patients weighing >35 kg
  Arms: Omeprazole

SUMMARY:
Crohn's disease (CD) is an inflammatory bowel disease characterized by chronic symptoms that include periods of exacerbation and remission. The exact cause of CD is not fully understood, but it is believed to result from a combination of genetic predispositions, immunological disorders, and environmental factors. The incidence of CD is on the rise, particularly among children, with estimates suggesting that it affects 1 in 500 people in Western Europe and North America. Notably, one in four patients diagnosed with CD are children. The inflammatory changes associated with CD can affect the entire thickness of the gastrointestinal wall and can occur anywhere along the gastrointestinal tract, from the mouth to the anus. Persistent inflammation in the gastrointestinal tract increases the risk of cancer, which is already heightened in patients with CD. In the pediatric population, inflammation in the esophagus, stomach, and duodenum is present in about 30% of cases and is associated with a poorer prognosis. Another factor linked to a worse prognosis is the age at diagnosis; younger patients tend to have a more severe disease course. Therefore, all children with CD generally experience a worse prognosis compared to adults. The treatment of CD is life-lasting and often challenging. It includes dietary modifications, pharmacological interventions, and sometimes surgical procedures, depending on the disease's activity and the location of the inflammation. The pharmacological treatment typically involves several types of medications: 5-ASA preparations, immunomodulatory drugs, biological drugs and local treatments such as suppositories, enemas and prolonged-release capsules. The most effective treatment approaches combine both systemic and local medications targeted at the affected areas of the intestine. In local treatment for CD, budesonide plays a crucial role. This corticosteroid has a strong anti-inflammatory effect and is characterized by low bioavailability, with 90% of the drug metabolized in the liver. Consequently, only 10% reaches the systemic circulation, minimizing the potential for adverse effects. Currently, budesonide is used to treat inflammatory changes in the distal small intestine (via sustained-release or enteric-coated capsules), rectum, and sigmoid colon (as rectal foam), or in the large intestine (with multimatrix tablets). Unfortunately, there is no local treatment available for patients with CD who have inflammation in the esophagus, stomach, or duodenum. Recommendations often suggest the use of antacids, such as proton pump inhibitors, which typically alleviate symptoms but do not promote remission of the inflammation. Given this gap in treatment, it has been hypothesized that adding locally acting budesonide to systemic therapy could be effective for children with inflammatory changes in the esophagus, stomach, and/or duodenum associated with CD. The aim of this study is to assess the efficacy of locally applied budesonide in treating these specific inflammatory changes in pediatric patients with Crohn's disease.

DETAILED DESCRIPTION:
The prospective, randomized, single-blind study. Children with CD who meet the inclusion criteria will be randomly assigned, based on a computer-generated randomization list, to one of two groups. One group will be treated with budesonide and the other with omeprazole. All preparations will be taken orally by children every 12 hours for 8 weeks. The child will swallow the capsule/capsules (with omeprazole) with water or the content of the ampoule/ampoules (budesonide). For 30 minutes after swallowing each dose, the patient will not drink, eat, chew gum or brush their teeth. After 30 minutes, the patient will be asked to rinse their mouth. The expected time from the start of screening to randomization is 2 weeks. Follow-up visits will take place at weeks 4, 8, and 12 of the study. The permitted deviation from the designated checkpoints (including randomization) is +/- 4 days. At the visit after 8 weeks, a control gastroscopy will be performed with collection of samples for histopathological evaluation. The 12-week visit will be a follow-up check

ELIGIBILITY:
Inclusion Criteria:

* CD diagnosed according to the commonly accepted Porto criteria, which take into account clinical, endoscopic and histopathological criteria;
* inflammatory changes in the esophagus and/or stomach and/or duodenum found in the endoscopic examination (assessed by 2 independent endoscopists) and confirmed in the histopathological examination (in the Paris scale, CD activity: L4a, i.e. involvement of the upper gastrointestinal tract up to the ligament of Treitz);
* stable, understood as no treatment modification, CD treatment for ≥2 weeks.

Exclusion Criteria:

* other than CD, causes of inflammatory changes in the esophagus and/or stomach and/or duodenum such as: reflux esophagitis, herpetic esophagitis, cytomegalovirus esophagitis, eosinophilic esophagitis and/or gastritis and/or duodenitis, Helicobacter pylori infection;
* use of systemic steroids for up to 30 days before enrollment in the study;
* use of inhaled steroids for up to 30 days before enrollment in the study;
* use of IPP for up to 30 days before enrollment in the study;
* acute viral or bacterial infection for up to 30 days before enrollment in the study;
* morning cortisol <5 ug/dl;
* lack of informed consent from the child's parents or guardians to participate in the study; in the case of children ≥16 years of age, lack of the child's consent to participate in the study.
* pregnancy
* breastfeeding;
* lack of consent of a woman of childbearing age or a fertile man to follow contraceptive recommendations during the study;
* history of cancer in the patient.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 8 weeks
  the percentage of patients with no endoscopic and histopathological changes in the esophagus, stomach and duodenum

SECONDARY OUTCOMES:
Endoscopic effectiveness | 8 weeks
  the percentage of patients with no endoscopic changes in the esophagus, stomach and duodenum, respectively (which were present at the time of study entry)
Histopathological effectiveness | 8 weeks
  the percentage of patients with no histopathological changes in the esophagus, stomach and duodenum, respectively
Disease activity | 8 weeks
  disease activity assessed on the Pediatric Crohn Disease Activity Index scale
Symptoms resolution | 4, 8 and 12 week
  the percentage of patients who had resolution of upper gastrointestinal symptoms
Adverse reactions | 4, 8 and 12 week
  the percentage of patients with adverse steroid reactions
Toleranc | 4 and 8 week
  treatment tolerance assessment on a 10-point VAS scale

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - Jagiellonian University, Krakow
  - Poznań University of Medical Sciences, Poznan
  - Medical University of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: No